CLINICAL TRIAL: NCT00000921
Title: A Phase II, Randomized, Placebo-Controlled Study of the Immunologic and Virologic Effects of Prednisone on HIV-1 Infection
Brief Title: The Effects of Prednisone on HIV Levels and the Immune System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 349
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Prednisone; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Prednisone

INTERVENTIONS:
Drug: Prednisone

SUMMARY:
The purpose of this study is to see if it is safe and effective to give prednisone to HIV-infected patients.

Prednisone is a corticosteroid, a hormone produced by the body that inhibits immune cell responses. Prednisone may be able to lower the level of HIV in the body (viral load) by reducing the number of cells that HIV can infect. At the same time, prednisone may be able to increase CD4 cell counts (cells of the immune system that fight infection).

DETAILED DESCRIPTION:
By inhibiting cellular activation, corticosteroids such as prednisone may inhibit HIV expression and reduce the population of potentially infectable cells. Furthermore, no studies have been performed to systematically evaluate immune function in prednisone-treated, HIV-infected patients or the immune mechanisms that may facilitate increases in CD4+ cell number. This study explores this issue.

Patients are separated into 2 arms according to whether or not they are currently receiving a protease inhibitor (PI) as part of their antiretroviral (ARV) therapy regimen (PI vs no PI therapy). Arm I: Current stable ARV therapy plus prednisone for 8 weeks, followed by 4 weeks at half the prior dose, then a 2-week taper. Arm II: Current stable ARV therapy plus prednisone placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 cell count of 200-600 cells/mm3 within 30 days of study entry. (This study has been changed. You now must have a CD4 cell count of 200-700 cells/mm3 within 45 days of study entry.)
* Have had your viral load measured within 30 days of study entry.
* Have been on stable anti-HIV therapy with at least two anti-HIV agents for at least 12 weeks, and you intend to remain on this therapy during the study.
* Are at least 18 years of age.
* Agree to abstain from sex or use effective methods of birth control during the study and for 30 days after.

Exclusion Criteria

You will not be eligible for this study if you:

* Abuse alcohol or drugs or have a serious psychological condition.
* Are allergic to prednisone or other corticosteroids.
* Have a history of opportunistic (AIDS-related) infections, including cytomegalovirus (CMV), Mycobacterium avium complex (MAC), or Kaposi's sarcoma (KS).
* Have a history of a serious medical condition, including heart problems, tuberculosis (TB), cancer, diabetes, or osteoporosis.
* Are being treated for herpes at study entry.
* Have received certain medications, including blood pressure medication.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118
Dates: Start 1996-08; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wallis R, Study Chair; Jacobson J, Study Chair; Kalayjian R, Study Chair
Locations (18):
- United States (18):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii / Leahi Hosp, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Wallis RS, Kalayjian R, Jacobson JM, Fox L, Purdue L, Shikuma CM, Arakaki R, Snyder S, Coombs RW, Bosch RJ, Spritzler J, Chernoff M, Aga E, Myers L, Schock B, Lederman MM. A study of the immunology, virology, and safety of prednisone in HIV-1-infected subjects with CD4 cell counts of 200 to 700 mm(-3). J Acquir Immune Defic Syndr. 2003 Mar 1;32(3):281-6. doi: 10.1097/00126334-200303010-00006. PMID 12626887